CLINICAL TRIAL: NCT03305471
Title: A Phase 1b Study, to Assess the Safety, Tolerability, Pharmacodynamics, and Pharmacokinetics of Repeated Doses of DS-2330b Alone and When Co-administered With Sevelamer in Patients on Chronic Hemodialysis
Brief Title: DS2330b Alone and With Sevelamer in Patients on Chronic Hemodialysis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DS2330-A-U103
Record Dates: First submitted 2017-10-04; First posted 2017-10-10 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Hyperphosphatemia
Keywords: Chronic hemodialysis; Investigational drug
MeSH Terms: conditions — Hyperphosphatemia | interventions — Sevelamer

STUDY DESIGN:
Intervention Model Description: Part A has a 2-period, open-label, randomized, 2-way crossover design with a single dose of Treatments A1 and A2
  Part B participants are randomized with a 2:3:3:3 ratio to Treatment B1, B2, B3, and B4, respectively, using a double-blind, repeated dose, parallel design
  Part C is an optional, single-arm, open label, repeated dose design
Who Masked: Participant, Investigator
Masking Description: Masking description is for Part B only - Parts A and C are Open Label, so have no masking
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Part A: DS-2330b PIB, then Tablet (Experimental): On a non-dialysis day, participants are given a single 250 mg dose of DS-2330b PIB [Treatment A1] right after breakfast. At least 3 days will be allowed to let the first dose wash out. Then on a non-dialysis day the participants are given a single 250 mg dose of DS-2330b in tablet form [Treatment A2] right after breakfast.
  Interventions: Drug: DS-2330b PIB; Drug: DS-2330b Tablet
- Part A: DS-2330b Tablet, then PIB (Experimental): On a non-dialysis day, participants are given a single 250 mg dose of DS-2330b in tablet form [Treatment A2] right after breakfast. At least 3 days will be allowed to let the first dose wash out. Then on a non-dialysis day the participants are given a single 250 mg dose of DS-2330b PIB [Treatment A1] right after breakfast.
  Interventions: Drug: DS-2330b PIB; Drug: DS-2330b Tablet
- Part B: Placebo (Placebo Comparator): Participants are given placebo three times daily [Treatment B1]
  Interventions: Drug: Placebo
- Part B: DS-2330b PIB (Experimental): Participants are given 400 mg of DS-2330b PIB three times daily [Treatment B2]
  Interventions: Drug: DS-2330b PIB
- Part B: DS-2330b PIB + Sevelamer (Experimental): Participants are given 400 mg of DS-2330b PIB along with 1.6 grams of sevelamer three times daily [Treatment B3]
  Interventions: Drug: DS-2330b PIB; Drug: Sevelamer
- Part B: Placebo + Sevelamer (Experimental): Participants are given placebo along with 1.6 grams of sevelamer three times daily [Treatment B4]
  Interventions: Drug: Placebo; Drug: Sevelamer
- Part C: DS-2330b Tablet + Sevelamer (Experimental): Participants are given one 250 mg dose of DS-2330b in tablet form along with 1.6 grams of sevelamer three times daily [Treatment C]
  Interventions: Drug: Sevelamer; Drug: DS-2330b Tablet

INTERVENTIONS:
Drug: DS-2330b PIB — DS-2330b as powder in bottle with stock solution (PIB)
  Arms: Part A: DS-2330b PIB, then Tablet; Part A: DS-2330b Tablet, then PIB; Part B: DS-2330b PIB; Part B: DS-2330b PIB + Sevelamer
Drug: Placebo — Placebo matching stock solution in bottle
  Arms: Part B: Placebo; Part B: Placebo + Sevelamer
Drug: Sevelamer — Sevelamer is a phosphate binder. It is used to decrease serum phosphate (Pi) level in people with chronic kidney disease who are on dialysis.
  Other Names: Sevelamer carbonate
  Arms: Part B: DS-2330b PIB + Sevelamer; Part B: Placebo + Sevelamer; Part C: DS-2330b Tablet + Sevelamer
Drug: DS-2330b Tablet — DS-2330b as tablet formulation
  Arms: Part A: DS-2330b PIB, then Tablet; Part A: DS-2330b Tablet, then PIB; Part C: DS-2330b Tablet + Sevelamer

SUMMARY:
This three-part study will be performed with participants on chronic hemodialysis.

* Part A will assess plasma pharmacokinetics of DS2330a (free form of DS2330b) after a single dose of powder in bottle (PIB) or tablet formulations of DS2330b
* Part B will test the safety, tolerability, and effects on serum phosphate (Pi) of 14-day repeated oral doses of DS-2330b PIB when given alone and when given along with sevelamer carbonate three times a day
* Part C is optional, and will test the effects on serum phosphate (Pi) of 14-day repeated oral doses of DS-2330b tablets when given with sevelamer carbonate

After screening, participants should expect the study to last about 21 days for Part A, and 46 days for Parts B and C.

ELIGIBILITY:
Inclusion Criteria:

* Has a body mass index (BMI) of 18 kg/m^2 to 40 kg/m^2 (inclusive)
* Is on prescribed maintenance hemodialysis (three times a week) for at least 3 months before Screening with adequacy demonstrated by a dialysis clearance within 3 months before the first dose of the investigational medicinal product
* Has permanent vascular access [arteriovenous (A-V) fistula or graft]
* Is willing to comply with protocol-specified methods for family planning
* For Parts B and C only:

  1. Has protocol-specified acceptable serum Pi levels at Screening and in serum Pi after up to 3 weeks of washout from all Pi binders
  2. Has protocol-specified acceptable serum Ca^2+ level and intact parathyroid hormone (iPTH) level at screening

Exclusion Criteria:

* Is employed by the clinic or the sponsor
* Has family relationship with another study participant
* Has any history, current condition, or drug use that per protocol or in the opinion of the investigator might compromise:

  1. safety of the participant or their children
  2. safety of study staff
  3. analysis of study results
* For Parts B and C only:

  1. Is not able to take sevelamer carbonate
  2. Has had partial or total parathyroidectomy within the last six months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-08-17 (Actual); Primary Completion 2019-01-03 (Actual); Study Completion 2019-01-03 (Actual)

PRIMARY OUTCOMES:
Part A, Period 1: Maximum concentration (Cmax) of DS-2330a | Period 1, Pre-dose to 48 hours post-dose
Part A, Period 2: Cmax of DS-2330a | Period 2, Pre-dose to 48 hours post-dose
Part A, Period 1: Time to maximum concentration (Tmax) of DS-2330a | Period 1, Pre-dose to 48 hours post-dose
Part A, Period 2: Tmax of DS-2330a | Period 2, Pre-dose to 48 hours post-dose
Part A, Period 1: Area under the drug concentration curve (AUC) for DS-2330a over 24 hours (AUC-24) | Period 1, Pre-dose to 24 hours post-dose
Part A, Period 2: AUC for DS-2330a for DS-2330a over 24 hours (AUC-24) | Period 2, Pre-dose to 24 hours post-dose
Part A, Period 1: AUC at the last observable concentration (AUClast) and to infinity (AUCinf) for DS-2330a | Period 1, Pre-dose to 48 hours post-dose
  Categories (with the same unit of measure ng*hr/mL): AUClast, AUCinf
Part A, Period 2: AUClast and AUCinf for DS-2330a | Period 2, Pre-dose to 48 hours post-dose
  Categories (with the same unit of measure ng*hr/mL): AUClast, AUCinf
Parts B and C: Serum phosphate (Pi) levels before hemodialysis | within 15 days
All Parts: Number of trial participants with treatment-emergent adverse events (TEAEs) | through trial completion (about 15 months)
  TEAEs are adverse events (side effects) associated with taking an investigational product, whether or not they were caused by the investigational product. Clinically significant changes in physical exam findings, vital signs, electrocardiograms, clinical lab tests and thyroid function are recorded as TEAEs.

SECONDARY OUTCOMES:
Parts B and C: Cmax of DS-2330a | within 24 hours on Day 1
Parts B and C: Cmax of DS-2330a | within 24 hours on Day 13
Parts B and C: Tmax of DS-2330a | within 24 hours, Day 1
Parts B and C: Tmax of DS-2330a | within 24 hours, Day 13
Parts B and C: AUC-24 for DS-2330a | Day 1
Parts B and C: AUC-24 for DS-2330a | Day 13
Parts B and C: AUCinf for DS-2330a | Day 1
Parts B and C: AUCinf for DS-2330a | Day 13
Parts B and C: Minimum concentration (Ctrough) of DS-2330a | within 11 days
  Trough blood levels for DS-2330a will be collected before the morning dose (prior to breakfast)
Part B: Dialysis clearance of DS-2330a | on Day 11

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (4):
- United States (4):
  - DaVita Clinical Research, Lakewood, Colorado
  - Orlando Clinical Research Center, Orlando, Florida
  - DaVita Clinical Research, Minneapolis, Minnesota
  - Prism Clinical Research, Saint Paul, Minnesota

REFERENCES:
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086